CLINICAL TRIAL: NCT04961983
Title: A Comprehensive Travel Health Education Improving Attitude, Subjective Norm, Perceived Behavioral Control, Role Identity, Actual Behavioral Control, and Intention to Provide Travel Health Information of Tour Guides in Bali
Brief Title: A Comprehensive Travel Health Education for Tour Guides in Bali, Indonesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Ni Made Sri Nopiyani, MD, MPH, Udayana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021.03.1.0515
Record Dates: First submitted 2021-07-09; First posted 2021-07-14 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Behavior, Health; Travel-Related Illness
Keywords: travel health; health promotion; tour guides
MeSH Terms: conditions — Health Behavior; Travel-Related Illness

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to two groups (intervention and control groups) in parallel for the duration of the study. The allocation of participants into the intervention and control groups will be carried out using permuted block randomization technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Tour guides who will receive a comprehensive travel health education model.
  Interventions: Behavioral: Comprehensive Travel Health Education Model
- Control group (No Intervention): Tour guides who will receive no intervention.

INTERVENTIONS:
Behavioral: Comprehensive Travel Health Education Model — The comprehensive travel health education model consists of:
  1. Online training: 10 hours (2 days) online education via Zoom. The topics that will be delivered during the training includes:
     * The potential roles of tour guides in tourists' health,
     * The importance of travel health information for tourists,
     * Assessment of tourist's health risks,
     * Prevention and first aid of various travel health problems Topics related to tour guides will be delivered by the tourism experts, while topics related to travel health will be provided by travel medicine experts, Faculty of Medicine, Udayana University. Participants will also receive a travel health guide book.
  2. Weekly travel health Information sharing through WhatsApp group for 2 months.
  Arms: Intervention group

SUMMARY:
This is a field trial with a randomized pre-test post-test control group design. This trial is the second phase of an exploratory mixed methods research. Prior to this trial, a qualitative study through in-depth interviews to tour guides from 11 language divisions and also policy makers of Indonesian Tour Guide Association Bali branch (HPI Bali). The education model for tour guides were developed based on the integration of theory of planned behavior (TPB) and identity theory. This educational model is expected to improve the behavior of tour guides in providing travel health information to tourists they serve, which is currently still lacking. However, due to the COVID-19 pandemic, the measurement of behavior can not be conducted. Therefore, this trial aims to test the efficacy of the comprehensive education model to improve the indirect and direct determinants of the behavior namely attitude, subjective norms, perceived behavioral control, role identity, actual behavioral control and behavioral intention.

The research hypothesis are:

1. The comprehensive travel health education model improves the attitude of tour guides towards providing travel health information to tourists?
2. The comprehensive travel health education model improves the subjective norms of tour guides towards providing travel health information to tourists?
3. The comprehensive travel health education model improves the perceived behavioral control of tour guides in providing travel health information to tourists?
4. The comprehensive travel health education model improves the role identity of tour guides as a travel health promoter for tourists?
5. The comprehensive travel health education model improves the actual behavioral control of tour guides in providing travel health information to tourists?
6. The comprehensive travel health education model improves the intention of tour guides to provide travel health information to tourists?

DETAILED DESCRIPTION:
1. Study design: This is a field trial with a randomized pre-test post-test control group design. This trial is the second phase of an exploratory mixed methods research.
2. Study setting: Data collection will be conducted in Bali, Indonesia, started from September 2021 to February 2022.
3. Study population: The target population in this study are all general tour guides in Bali, Indonesia. The accessible population are general tour guides who are registered as members of HPI Bali who can be reached during the data collection period.
4. Sample size: The calculation of the minimum sample size in this study was carried out with the assistance of the WHO Sample Size Determination software using the hypothesis test formula for the mean difference of two populations (one-sided).

   Based on the sample size calculation with the above formula, the minimum sample size for each group is 69 tour guides. Taking into account the drop-out rate of 10%, the number of samples for each group is 76 tour guides. Thus, the total number of samples for intervention and comparison groups in this study is 152 tour guides.
5. Sample selection: The sample selection was carried out with disproportionate stratified random sampling using a sampling frame namely the list of tour guides who are registered as the members of Indonesian Guides Association (HPI) Bali Branch from 11 language divisions. The number of samples in each division for intervention and control group ranged from 5 to 8 subjects.
6. Sample allocation: Permuted block randomization.
7. Study variables:

   1. Dependent variable is comprehensive travel health education model.
   2. Intermediate variables are:

      * attitude towards providing travel health information to tourists,
      * subjective norms towards providing travel health information to tourists,
      * perceived behavioral control of providing travel health information to tourists,
      * role identity,
      * actual behavioral control.
   3. Dependent variable is intention to provide travel health information to tourists.
   4. Controll variables are:

   Controlled by design:
   * history of formal health education,
   * ownership of a smartphone or laptop with WhatsApp and Zoom application,
   * familiarity with Zoom usage,
   * familiarity with WhatsApp usage.

   Controlled by analysis:
   * age,
   * sex,
   * education,
   * length of work,
   * employment status,
   * tourists' country of origin,
   * type of tourism activities,
   * employer's policy.
8. Research instrument:

The instrument that will be used in this study is a questionnaire. The measurement using questionnaire will be conducted before the intervention (pre-test) and after the intervention (post-test). The developed questionnaire consists of several parts, namely the identity or socio-demographic characteristics of the subjects, job characteristics, characteristics of tourists served, attitudes, subjective norms, perceived behavioral control, role identity, actual behavior control and behavioral intentions.

The questionnaire was developed based on the guidelines for developing a questionnaire for TPB-based interventions and the results of the qualitative study. The assessment for each statement item on the attitude, subjective norm, perceived behavioral control and role identity, uses a Likert scale consisting of seven scales, namely: 1 = strongly disagree, 2 = disagree; 3 = disagree, 4 = undecided, 5 = somewhat agree, 6 = agree; 7 = strongly agree.

The questionnaire on the actual behavior control section consists of questions related to knowledge about prevention and first aid for tourism health problems. Questions to measure knowledge were developed based on the material provided during the intervention. The correct answer for each knowledge question will get a score 1, while the wrong or 'do not know' answer will be given a score 0.

The questionnaire on the behavioral intention section is also written in statement format. The assessment for each statement item uses a Likert scale consisting of seven scales, namely: a scale of 1 = strongly not intending, 2 = not intending; 3 = lack of intention, 4 = undecided, 5 = somewhat intend, 6 = intend; 7 = very intent.

The validity and reliability of the questionnaire will be tested before it being used in data collection. Twenty tour guides will be involved in the pilot test of the questionnaire. If necessary, improvements will be made to the questionnaire based on the test results. The questionnaire is self-administered and will be given to the subjects in digital format.

9. Data analysis:

1. Descriptive statistic Quantitative data obtained from the questionnaire will be analyzed descriptively by calculating the frequency distribution for data on a categorical scale and by calculating the total value, mean, median, standard deviation and range of values from minimum to maximum on continuous scale data. On the variables of attitude, subjective norm, perceived behavioral control, and role identity, a positive statement will get a score of 1 = strongly disagree; 1 = strongly disagree; 2 = disagree; 3 = disagree; 4 = doubtful; 5 = somewhat agree; 6 = agree; 7 = strongly agree. As for negative statements, the score given is the opposite, namely a score of 7 = strongly disagree; 6 = disagree; 5 = disagree; 4 = doubtful; 3 = somewhat agree; 2 = agree; 1 = strongly agree. The actual behavioral control score was 1 for correct answer and 0 for wrong answer and 'do not know' answer.
2. Chi square test Comparison of sample characteristics in the intervention and control groups in terms of control variables (age, gender, education, length of work, employment status, tourists' country of origin, type of tourism activities and employer's policy) was also carried out using the chi square test. Through this test, it will be known whether there are differences in the two groups based on these variables. If the p value > 0.05, the two groups are the same (comparable), whereas if p value ≤ 0.05 then the two groups are different in terms of the variables tested. Variables that have a p value ≤ 0.05 will be tested in multivariate analysis.
3. Normality test Data normality test is conducted to determine whether or not the data on attitude, subjective norms, perceived behavioral control, actual behavior control, role identity and behavioral intentions scores are normally distributed, as a prerequisite for being able to perform parametric statistical tests. Based on the sample size, the normality test will be carried out using the Kolmogorov-Smirnov test. If the normality test produces a p value > 0.05 then the data distribution is normally distributed. On the other hand, the data is not normally distributed if the p ≤ 0.05.
4. Homogeneity test The purpose of the homogeneity test is to find out whether the two groups to be compared have the same variance. According to the sample size, homogeneity test will be carried out using Levene's test. If the results of the homogeneity test show a p value > 0.05 then the variance between groups is homogeneous. On the other hand, if the p value ≤ 0,05, the variance of the two groups is not homogeneous.
5. Mean comparison test The mean comparison test will be conducted to determine whether there is a difference in the mean between the intervention and the control group (difference in the mean of two independent samples). The mean comparison procedure used in this study is the independent samples t test. However, testing with independent samples t test is a parametric test which assumes the data is normally distributed and both groups have the same variance. The interpretation of the test results is that Ho is accepted if the p value > 0.05 or the zero value lies within the confidence interval for the difference in the mean, on the other hand Ho is rejected if the p value ≤ 0,05 or the zero value lies outside the confidence interval for the mean difference of the two groups. If the data is not normally distributed, the data will be transformed. Furthermore, if the transformation cannot make the data normally distributed, the data will be analyzed by non-parametric statistical tests, namely the Mann Whitney U test.

   In addition to the comparison of the mean between the intervention and comparison groups, a comparison test of the means was also carried out for the control variables. For categorical-scale control variables with two categories, a t-test was performed, such as a comparative analysis of the mean for the intervention and control groups. Meanwhile, for control variables that have more than two categories, an analysis of variance (ANOVA) test will be carried out. If the assumptions for the parametric statistical test are not met, the Kruskal-Wallis test is performed.
6. Multivariate analysis After the bivariate analysis, a multivariate analysis was carried out which aims to control the inter-correlation between the variables under study. In multivariate analysis, all dependent variables are tested simultaneously. If the assumptions for parametric statistical analysis are met, the statistical test used is multivariate analysis of variance (MANOVA). MANOVA is chosen because there is more than one continuous-scale dependent variable to be tested and more than one categorical-scale independent variable with two or more categories. If the assumptions are not met, then a non-parametric MANOVA statistical test is performed.

ELIGIBILITY:
Inclusion Criteria:

1. Active members of HPI Bali,
2. Age less than 55 years old,
3. Have worked as a tour guide for one year or more,
4. Have a smart phone or laptop that equipped with Zoom and WhatsApp application,
5. Familiar with Zoom meeting,
6. Using WhatsApp actively.

Exclusion Criteria:

1. Holding a structural position at HPI Bali,
2. Unwilling to work as a tour guide after the re-opening of tourism,
3. Have a formal health education background,
4. Unwilling to participate in this study.

Ages: 20 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Mean score of attitude | 3 months
  Attitude is a psychological tendency expressed by tour guides towards the behavior of providing travel health information to tourists. Attitude will be measured through a self-administered questionnaire developed based on the TPB questionnaire development guideline. The data measurement scale is ordinal which is expressed on a Likert scale (1 = strongly disagree, 2 = disagree; 3 = disagree, 4 = neutral, 5 = somewhat agree, 6 = agree; 7 = strongly agree). Data will be analysed in interval scale.
Mean score of subjective norm | 3 months
  Subjective norm is the perception of tour guides on the extent to which the behavior of providing health information to tourists is a behavior that is expected by the tourists, by their employers, HPI, and the community. Subjective norms will be measured through a self-administered questionnaire which was developed based on TPB questionnaire development guideline. The measurement scale is ordinal which is expressed on a Likert scale (1 = strongly disagree, 2 = disagree; 3 = disagree, 4 = neutral, 5 = somewhat agree, 6 = agree; 7 = strongly agree). Data will be analysed in interval scale.
Mean score of perceived behavioral control | 3 months
  Perceived behavioral control is the confidence of tour guides in their ability to carry out the behavior of providing information to tourists regarding prevention and first aid of health problems. Perceived behavioral control will be measured through a self-administered questionnaire which was developed based on the TPB questionnaire development guideline. The measurement scale is ordinal which is expressed on a Likert scale (1 = strongly disagree, 2 = disagree; 3 = disagree, 4 = neutral, 5 = somewhat agree, 6 = agree; 7 = strongly agree). Data will be analysed in interval scale.
Mean score of actual behavioral control | 3 months
  Actual behavioral control is tour guide's knowledge about the prevention of travel health problems and first aid to tourists who experience health problems. Actual behavioral control will be measured through a self-administered questionnaire. The measurement scale is ordinal which is expressed on a Likert scale (1 = strongly disagree, 2 = disagree; 3 = disagree, 4 = neutral, 5 = somewhat agree, 6 = agree; 7 = strongly agree). Data will be analysed in interval scale. Knowledge measurement scale is interval. The correct answer for each knowledge question will get a score = 1, while the question with the wrong answer or do not know gets a score = 0. Data will be analysed in interval scale.
Mean score of role identity | 3 months
  Role identity is tour guide's perception of the extent to which the provision of information related to the prevention and first aid of tourism health problems to tourists is a part of the tour guide's role. Role identity will be measured through a self-administered questionnaire.The measurement scale is ordinal which is expressed on a Likert scale (1 = strongly disagree, 2 = disagree; 3 = disagree, 4 = neutral, 5 = somewhat agree, 6 = agree; 7 = strongly agree). Data will be analysed in interval scale.
Mean score of behavioral intention | 3 months
  Behavioral intention is the willingness of tour guides to convey information related to the prevention and first aid of travel health problems to the tourists they serve. Intention will be measured through a self-administered questionnaire which was developed based on the TPB questionnaire development guideline. The data measurement scale is ordinal which is expressed on a Likert scale (1 = strongly disinterested, 2 = not intending; 3 = lack of intention, 4 = neutral, 5 = somewhat intend, 6 = intend; 7 = very intend). Data will be analysed in interval scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ni Made Sri Nopiyani, MD, MPH, Principal Investigator — Udayana University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ajzen I. The theory of planned behaviour: reactions and reflections. Psychol Health. 2011 Sep;26(9):1113-27. doi: 10.1080/08870446.2011.613995. PMID 21929476
- [Background] Ajzen I. The theory of planned behaviour is alive and well, and not ready to retire: a commentary on Sniehotta, Presseau, and Araujo-Soares. Health Psychol Rev. 2015;9(2):131-7. doi: 10.1080/17437199.2014.883474. Epub 2014 Feb 12. No abstract available. PMID 26209198
- [Background] Alqahtani AS, Tashani M, Heywood AE, Booy R, Rashid H, Wiley KE. Exploring Australian Hajj Tour Operators' Knowledge and Practices Regarding Pilgrims' Health Risks: A Qualitative Study. JMIR Public Health Surveill. 2019 May 23;5(2):e10960. doi: 10.2196/10960. PMID 31124464
- [Background] Johansson Arhem KM, Gysin N, Nielsen HV, Surya A, Hellgren U. Low and Declining Risk for Malaria in Visitors to Indonesia: A Review of Local Indonesian and European Travelers' Data and a Suggestion for New Prophylactic Guidelines. J Travel Med. 2015 Nov-Dec;22(6):389-95. doi: 10.1111/jtm.12233. Epub 2015 Oct 13. PMID 26464104
- [Background] Armitage CJ, Conner M. Efficacy of the Theory of Planned Behaviour: a meta-analytic review. Br J Soc Psychol. 2001 Dec;40(Pt 4):471-99. doi: 10.1348/014466601164939. PMID 11795063
- [Background] Avcikurt C, Koroglu O, Koroglu A, Avcikurt AS. HIV/AIDS awareness and attitudes of tour guides in Turkey. Cult Health Sex. 2011 Feb;13(2):233-43. doi: 10.1080/13691058.2010.522733. PMID 21058083
- [Background] Bauer I. The health impact of tourism on local and indigenous populations in resource-poor countries. Travel Med Infect Dis. 2008 Sep;6(5):276-91. doi: 10.1016/j.tmaid.2008.05.005. Epub 2008 Aug 9. PMID 18760250
- [Background] Bertman V, Petracca F, Makunike-Chikwinya B, Jonga A, Dupwa B, Jenami N, Nartker A, Wall L, Reason L, Kundhlande P, Downer A. Health worker text messaging for blended learning, peer support, and mentoring in pediatric and adolescent HIV/AIDS care: a case study in Zimbabwe. Hum Resour Health. 2019 Jun 7;17(1):41. doi: 10.1186/s12960-019-0364-6. PMID 31174543
- [Background] Broglio K. Randomization in Clinical Trials: Permuted Blocks and Stratification. JAMA. 2018 Jun 5;319(21):2223-2224. doi: 10.1001/jama.2018.6360. No abstract available. PMID 29872845
- [Background] Cooke R, Dahdah M, Norman P, French DP. How well does the theory of planned behaviour predict alcohol consumption? A systematic review and meta-analysis. Health Psychol Rev. 2016 Jun;10(2):148-67. doi: 10.1080/17437199.2014.947547. Epub 2014 Sep 17. PMID 25089611
- [Background] Dunleavy G, Nikolaou CK, Nifakos S, Atun R, Law GCY, Tudor Car L. Mobile Digital Education for Health Professions: Systematic Review and Meta-Analysis by the Digital Health Education Collaboration. J Med Internet Res. 2019 Feb 12;21(2):e12937. doi: 10.2196/12937. PMID 30747711
- [Background] Gautret P, Angelo KM, Asgeirsson H, Lalloo DG, Shaw M, Schwartz E, Libman M, Kain KC, Piyaphanee W, Murphy H, Leder K, Vincelette J, Jensenius M, Waggoner J, Leung D, Borwein S, Blumberg L, Schlagenhauf P, Barnett ED, Hamer DH; GeoSentinel Global Surveillance Network. Rabies post-exposure prophylaxis started during or after travel: A GeoSentinel analysis. PLoS Negl Trop Dis. 2018 Nov 13;12(11):e0006951. doi: 10.1371/journal.pntd.0006951. eCollection 2018 Nov. PMID 30422981
- [Background] Giovanetti F. Methanol poisoning among travellers to Indonesia. Travel Med Infect Dis. 2013 May-Jun;11(3):190-3. doi: 10.1016/j.tmaid.2013.03.013. Epub 2013 Apr 6. PMID 23566856
- [Background] Grech V, Grech P, Fabri S. A risk balancing act - Tourism competition using health leverage in the COVID-19 era. Int J Risk Saf Med. 2020;31(3):121-130. doi: 10.3233/JRS-200042. PMID 32597822
- [Background] Hirata K, Ogawa T, Fujikura H, Ogawa Y, Hirai N, Nakagawa-Onishi T, Uno K, Takeyama M, Kasahara K, Nakamura-Uchiyama F, Konishi M, Mikasa K. Characteristics of health problems in returned overseas travelers at a tertiary teaching hospital in a suburban area in Japan. J Infect Chemother. 2018 Aug;24(8):682-685. doi: 10.1016/j.jiac.2018.02.003. Epub 2018 Mar 2. PMID 29503227
- [Background] Horvath LL, Murray CK, DuPont HL. Travel health information at commercial travel websites. J Travel Med. 2003 Sep-Oct;10(5):272-8. doi: 10.2310/7060.2003.2699. PMID 14531980
- [Background] Hsu SH, Huang HL, Lu CW, Cheng SY, Lee LT, Chiu TY, Huang KC. Tour leaders with detailed knowledge of travel-related diseases play a key role in disease prevention. Medicine (Baltimore). 2018 Feb;97(6):e9806. doi: 10.1097/MD.0000000000009806. PMID 29419678
- [Background] Ivatts SL, Plant AJ, Condon RJ. Travel health: perceptions and practices of travel consultants. J Travel Med. 1999 Jun;6(2):76-80. doi: 10.1111/j.1708-8305.1999.tb00836.x. PMID 10381958
- [Background] Kemp N, Grieve R. Face-to-face or face-to-screen? Undergraduates' opinions and test performance in classroom vs. online learning. Front Psychol. 2014 Nov 12;5:1278. doi: 10.3389/fpsyg.2014.01278. eCollection 2014. PMID 25429276
- [Background] Kolars JC. Rules of the road: a consumer's guide for travelers seeking health care in foreign lands. J Travel Med. 2002 Jul-Aug;9(4):198-201. doi: 10.2310/7060.2002.24042. No abstract available. PMID 12962614
- [Background] Kwong JC, Druce JD, Leder K. Zika virus infection acquired during brief travel to Indonesia. Am J Trop Med Hyg. 2013 Sep;89(3):516-7. doi: 10.4269/ajtmh.13-0029. Epub 2013 Jul 22. PMID 23878182
- [Background] Leder K, Borwein S, Chanthavanich P, Chatterjee S, Htun K, Marma ASP, Nakatani I, Ok JJ, Pakasi L, Pandey P, Piyaphanee W, Rupali P, Schwartz E, Shinozuka T, Phu PTH, Watanabe H, Visser J, Wilder-Smith A, Zhang M, McGuinness SL. Travel medicine perspectives of select travel medicine experts practicing in the Asia-Pacific region. J Travel Med. 2017 Jul 1;24(4). doi: 10.1093/jtm/tax012. No abstract available. PMID 28426112
- [Background] Leggat PA, Zwar NA, Hudson BJ; Travel Health Advisory Group, Australia. Hepatitis B risks and immunisation coverage amongst Australians travelling to southeast Asia and east Asia. Travel Med Infect Dis. 2009 Nov;7(6):344-9. doi: 10.1016/j.tmaid.2009.03.008. Epub 2009 May 9. PMID 19945011
- [Background] Lestelle C, Aymeric S, Maakaroun-Vermesse Z, Pouliquen A, Bernard L, Chandenier J, Grammatico-Guillon L. Impact of advice given to travelers concerning the main infectious risks associated with traveling in the tropics. Med Mal Infect. 2015 Jun;45(6):222-8. doi: 10.1016/j.medmal.2015.04.007. Epub 2015 May 27. PMID 26026227
- [Background] Liu Q, Peng W, Zhang F, Hu R, Li Y, Yan W. The Effectiveness of Blended Learning in Health Professions: Systematic Review and Meta-Analysis. J Med Internet Res. 2016 Jan 4;18(1):e2. doi: 10.2196/jmir.4807. PMID 26729058
- [Background] MacDougall LA, Gyorkos TW, Leffondre K, Abrahamowicz M, Tessier D, Ward BJ, MacLean JD. Increasing referral of at-risk travelers to travel health clinics: evaluation of a health promotion intervention targeted to travel agents. J Travel Med. 2001 Sep-Oct;8(5):232-42. doi: 10.2310/7060.2001.24016. PMID 11703905
- [Background] MacIntyre CR, Karki S, Sheikh M, Zwar N, Heywood AE. The role of travel in measles outbreaks in Australia - An enhanced surveillance study. Vaccine. 2016 Aug 17;34(37):4386-91. doi: 10.1016/j.vaccine.2016.07.023. Epub 2016 Jul 19. PMID 27449078
- [Background] Marchand C, Merrina F, Gagnayre R, Bouchaud O. A descriptive study of advising practices during travel health consultations in France. J Travel Med. 2017 Sep 1;24(5). doi: 10.1093/jtm/tax042. PMID 28931133
- [Background] Masyeni S, Yohan B, Somia IKA, Myint KSA, Sasmono RT. Dengue infection in international travellers visiting Bali, Indonesia. J Travel Med. 2018 Aug 1;25(1):tay061. doi: 10.1093/jtm/tay061. PMID 30113689
- [Background] McDermott MS, Oliver M, Svenson A, Simnadis T, Beck EJ, Coltman T, Iverson D, Caputi P, Sharma R. The theory of planned behaviour and discrete food choices: a systematic review and meta-analysis. Int J Behav Nutr Phys Act. 2015 Dec 30;12:162. doi: 10.1186/s12966-015-0324-z. PMID 26715190
- [Background] Muller JM, Simonet AL, Binois R, Muggeo E, Bugnon P, Liet J, Duong M, Chavanet P, Piroth L. The respect of recommendations provided in an international travelers' medical service: far from the cup to the lips. J Travel Med. 2013 Mar-Apr;20(2):78-82. doi: 10.1111/j.1708-8305.2012.00675.x. Epub 2012 Nov 27. PMID 23464713
- [Background] Pavli A, Silvestros C, Patrinos S, Lymperi I, Maltezou HC. Pre-travel preparation practices among business travellers to tropical and subtropical destinations: results from the Athens International Airport Survey. Travel Med Infect Dis. 2014 Jul-Aug;12(4):364-9. doi: 10.1016/j.tmaid.2013.12.004. Epub 2013 Dec 24. PMID 24529745
- [Background] Peng Y, Wu X, Atkins S, Zwarentein M, Zhu M, Zhan XX, Zhang F, Ran P, Yan WR. Internet-based health education in China: a content analysis of websites. BMC Med Educ. 2014 Jan 27;14:16. doi: 10.1186/1472-6920-14-16. PMID 24467710
- [Background] Raby E, Dyer JR. Endemic (murine) typhus in returned travelers from Asia, a case series: clues to early diagnosis and comparison with dengue. Am J Trop Med Hyg. 2013 Apr;88(4):701-3. doi: 10.4269/ajtmh.12-0590. Epub 2013 Jan 28. No abstract available. PMID 23358638
- [Background] Rodriguez-Garcia R. The health-development link: travel as a public health issue. J Community Health. 2001 Apr;26(2):93-112. doi: 10.1023/a:1005225129295. PMID 11322757
- [Background] Rolling T, Muhlenpfordt M, Addo MM, Cramer JP, Vinnemeier CD. Pre-travel advice at a crossroad: Medical preparedness of travellers to South and Southeast-Asia - The Hamburg Airport Survey. Travel Med Infect Dis. 2017 Jul-Aug;18:41-45. doi: 10.1016/j.tmaid.2017.07.008. Epub 2017 Jul 18. PMID 28733254
- [Background] Rowe SL, Thevarajan I, Richards J, Gibney K, Simmons CP. The Rise of Imported Dengue Infections in Victoria, Australia, 2010(-)2016. Trop Med Infect Dis. 2018 Jan 21;3(1):9. doi: 10.3390/tropicalmed3010009. PMID 30274408
- [Background] Sniehotta FF, Presseau J, Araujo-Soares V. Time to retire the theory of planned behaviour. Health Psychol Rev. 2014;8(1):1-7. doi: 10.1080/17437199.2013.869710. Epub 2014 Jan 2. No abstract available. PMID 25053004
- [Background] Sohail A, McGuinness SL, Lightowler R, Leder K, Jomon B, Bain CA, Peleg AY. Spectrum of illness among returned Australian travellers from Bali, Indonesia: a 5-year retrospective observational study. Intern Med J. 2019 Jan;49(1):34-40. doi: 10.1111/imj.13993. PMID 29869360
- [Background] Steffen R, deBernardis C, Banos A. Travel epidemiology--a global perspective. Int J Antimicrob Agents. 2003 Feb;21(2):89-95. doi: 10.1016/s0924-8579(02)00293-5. PMID 12615369
- [Background] Tappe D, Nemecek A, Zipp F, Emmerich P, Gabriel M, Gunther S, Dobler G, Schmidt-Chanasit J, Stich A. Two laboratory-confirmed cases of Japanese encephalitis imported to Germany by travelers returning from Southeast Asia. J Clin Virol. 2012 Jul;54(3):282-5. doi: 10.1016/j.jcv.2012.03.004. Epub 2012 Mar 31. PMID 22465340
- [Background] Thomson CA, Gibbs RA, Giele C, Firth MJ, Effler PV. Health Seeking Behaviours and Knowledge of Infectious Disease Risks in Western Australian Travellers to Southeast Asian Destinations: An Airport Survey. Trop Med Infect Dis. 2016 Jul 18;1(1):3. doi: 10.3390/tropicalmed1010003. PMID 30270854
- [Background] Topa G, Moriano JA. Theory of planned behavior and smoking: meta-analysis and SEM model. Subst Abuse Rehabil. 2010 Dec 6;1:23-33. doi: 10.2147/SAR.S15168. eCollection 2010. PMID 24474850
- [Background] Wirawan IMA, Wirawan DN, Kurniasari NMD, Merati KTP. Travel agent and tour guide perceptions on travel health promotion in Bali. Health Promot Int. 2020 Feb 1;35(1):e43-e50. doi: 10.1093/heapro/day119. PMID 30668759
- [Background] Wirawan IMA, Putri WCWS, Kurniasari NMD, Mulyawan KH, Hendrayana MA, Suharlim C. Geo-mapping of hazards, risks, and travel health services in Bali: Results from the first stage of the integrated travel health surveillance and information system at destination (TravHeSID) project. Travel Med Infect Dis. 2020 Sep-Oct;37:101698. doi: 10.1016/j.tmaid.2020.101698. Epub 2020 Apr 28. PMID 32360324
- [Background] Zimmermann R, Hattendorf J, Blum J, Nuesch R, Hatz C. Risk perception of travelers to tropical and subtropical countries visiting a swiss travel health center. J Travel Med. 2013 Jan-Feb;20(1):3-10. doi: 10.1111/j.1708-8305.2012.00671.x. Epub 2012 Nov 26. PMID 23279224
- [Derived] Nopiyani NMS, Januraga PP, Wirawan IMA, Bakta IM. Comprehensive Travel Health Education for Tour Guides: Protocol for an Exploratory Sequential Mixed Methods Research. JMIR Res Protoc. 2022 May 23;11(5):e33840. doi: 10.2196/33840. PMID 35604754